CLINICAL TRIAL: NCT02761577
Title: A Prospective Study on Incidence and Prevention of Contrast-induced Nephropathy in Croatia With the Use of Standard Laboratory Measures and Novel Biomarkers
Brief Title: A Prospective Study on Incidence and Prevention of Contrast-induced Nephropathy in Croatia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Ana Vujaklija Brajkovic, M.D. PhD, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16012011
Record Dates: First submitted 2016-04-29; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Diseases; Contrast Media Reaction
Keywords: Acetylcysteine; Sodium Bicarbonate; Lipocalins; Creatinine; Blood Urea Nitrogen
MeSH Terms: conditions — Kidney Diseases | interventions — Sodium Bicarbonate; Acetylcysteine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): perorally 1500 ml water on the day of the procedure
- Sodium bicarbonate (Experimental): 3 mL/kg/hour IV (in vein) of Sodium bicarbonate, an hour prior to angiography and 1 mL/kg/hour, within six hours after angiography
  Interventions: Drug: Sodium bicarbonate
- N-acetylcysteine plus Sodium bicarbonate (Experimental): N-acetylcysteine (1200 mg twice a day, IV (in vein) ) one day before angiography, on the day of the angiography, and one day after the diagnostic procedure in addition to Sodium bicarbonate solution on the day of the angiography.
  Interventions: Drug: Sodium bicarbonate; Drug: N-acetylcysteine

INTERVENTIONS:
Drug: Sodium bicarbonate — 3 mL/kg/hour of Sodium bicarbonate, an hour prior to angiography and 1 mL/kg/hour, within six hours after angiography
  Other Names: NaHCO3
  Arms: N-acetylcysteine plus Sodium bicarbonate; Sodium bicarbonate
Drug: N-acetylcysteine — N-acetylcysteine (1200 mg twice a day, IV (in vein) ) one day before angiography, on the day of the angiography, and one day after the diagnostic procedure
  Other Names: fluimukan
  Arms: N-acetylcysteine plus Sodium bicarbonate

SUMMARY:
The study is analysis of the incidence of contrast-induced nephropathy (CIN) in patients with previously normal renal function undergoing angiography and comparison between the three different treatment protocols on renal function.

Patients are randomly assigned to the three groups: 1) peroral hydration, 2) Na bicarbonate (NaHCO3), and 3) NaHCO3 plus N-acetylcysteine (NAC) infusion.

Serum creatinine (SCr), blood urea nitrogen (BUN), and neutrophil gelatinase-associated lipocalin (NGAL) are measured before and 48 hours after the angiography. CIN was defined as an absolute increase of 0.5 mg/dL or a relative increase of >25% in creatinine levels 48-72 hours after the procedure

DETAILED DESCRIPTION:
Patients are randomly assigned to the three groups: 1) peroral hydration, 2) Na bicarbonate (NaHCO3), and 3) NaHCO3 plus N-acetylcysteine (NAC) infusion The first group of patients receives standard peroral hydration of 1500 ml water on the day of the procedure.

The second group receives 3 mL/kg/hour of Na bicarbonate, an hour prior to angiography and 1 mL/kg/hour, within six hours after angiography.

The third group receives parenteral NAC (1200 mg twice a day) one day before angiography, on the day of the angiography, and one day after the diagnostic procedure in addition to Na bicarbonate solution on the day of the angiography.

The low-osmolar iodinated contrast agent was used.

ELIGIBILITY:
Inclusion Criteria:

* angina (stable, unstable)
* coronary artery disease
* cardiomyopathy
* valvular disease
* vasculitis
* peripheral arterial disease

Exclusion Criteria:

* kidney dysfunction
* uncontrolled hypertension (systolic blood pressure >160 mm Hg and/or diastolic blood pressure >100 mm Hg)
* pregnancy
* lactation
* history of allergic reaction to contrast agents
* cardiogenic shock
* pulmonary edema
* multiple myeloma
* urgent coronary angiography
* receiving contrast agents two days prior to the study and 48 hours within the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
renal function before and after diagnostic procedure by measuring Serum creatinine in µmol/mL | 48 hours
  measure of serum creatinine before and after diagnostic procedure

SECONDARY OUTCOMES:
blood urea nitrogen in mmol/L | 48 hours
  measure of blood urea nitrogen before and after diagnostic procedure
neutrophil gelatinase-associated lipocalin in ng/mL | 48 hours
  measure of neutrophil gelatinase-associated lipocalin before and after diagnostic procedure

IPD SHARING:
Plan to Share IPD: Undecided